CLINICAL TRIAL: NCT07206810
Title: A Study of the Bortezomib, Lenalidomide, and Dexamethasone (VRD) Regimen for the Treatment of Newly Diagnosed Multiple Myeloma Patients
Brief Title: A Study of the Bortezomib, Lenalidomide, and Dexamethasone Regimen for the Treatment of Newly Diagnosed Multiple Myeloma Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: VRD-myeloma01
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Myeloma
Keywords: Newly diagnosed multiple myeloma; Lenalidomide; Bortezomib; Response; Survival
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Bortezomib, Lenalidomide, and Dexamethasone — In this study, transplant-eligible patients underwent autologous hematopoietic stem cell transplantation (auto-HSCT) after four cycles of VRD induction therapy, followed by two cycles of VRD consolidation therapy. Chemotherapy was administered in 28-day cycles as follows: subcutaneous bortezomib 1.3 mg/m² on days 1, 4, 8, and 11; oral lenalidomide 25 mg/day (or a dose-adjusted 10 mg based on renal function) from days 1 to 14; and intravenous dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11, and 12. Standard-risk patients received oral lenalidomide as maintenance therapy until disease progression. High-risk patients, defined as those with t(4;14), t(14;16), or del(17p), received bortezomib plus lenalidomide (V+R) as maintenance therapy until disease progression. Enrolled patients had complete clinical information at the time of initial diagnosis and received at least two cycles of VRD therapy.

SUMMARY:
A real-world prospective registry study for patients with newly diagnosed multiple myeloma (NDMM) has been conducted at the First Affiliated Hospital of Soochow University since August 2018. Diagnosis, staging, treatment response assessment, and risk stratification of MM were performed in accordance with the International Myeloma Working Group (IMWG) guidelines. In this study, transplant-eligible patients underwent autologous hematopoietic stem cell transplantation (auto-HSCT) after four cycles of VRD induction therapy, followed by two cycles of VRD consolidation therapy. Chemotherapy was administered in 28-day cycles as follows: subcutaneous bortezomib 1.3 mg/m² on days 1, 4, 8, and 11; oral lenalidomide 25 mg/day (or a dose-adjusted 10 mg based on renal function) from days 1 to 14; and intravenous dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11, and 12. Standard-risk patients received oral lenalidomide as maintenance therapy until disease progression. High-risk patients, defined as those with t(4;14), t(14;16), or del(17p), received bortezomib plus lenalidomide (V+R) as maintenance therapy until disease progression. Enrolled patients had complete clinical information at the time of initial diagnosis and received at least two cycles of VRD therapy. Frailty assessments were conducted prior to each chemotherapy cycle. The study protocol specified the following lenalidomide dosing based on renal function: patients with eGFR ≥60 ml/min/1.73 m² received oral lenalidomide 25 mg/day; those with 30 ml/min/1.73 m² ≤ eGFR < 60 ml/min/1.73 m² received oral lenalidomide 10 mg/day; and those with eGFR < 30 ml/min/1.73 m² or who were dialysis-dependent received oral lenalidomide 10 mg every other day. Long-term follow-up was performed to monitor treatment efficacy and survival status.

ELIGIBILITY:
Inclusion Criteria:

(1) diagnosis of active multiple myeloma according to the IMWG criteria; (2) age over 18 years; (3) newly diagnosed and treatment-naïve; (4) availability of complete clinical information; (5) receipt of at least two cycles of VRD regimen; and (6) regular follow-up at our department.

Exclusion Criteria:

(1) follow-up duration of less than 6 months; (2) incomplete clinical data; and (3) failure to receive regular treatment in our department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed multiple myeloma (NDMM) treated at the First Affiliated Hospital of Soochow University received the VRD regimen as induction therapy, followed by autologous hematopoietic stem cell transplantation (auto-HSCT) or non-transplantation management.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
response | before auto-HSCT
  sCR, CR, VGPR, PR, SD, PD

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No